CLINICAL TRIAL: NCT03632954
Title: Use of Cytal® Wound Matrix and MicroMatrix® for the Management of Wounds
Brief Title: Cytal® Wound Matrix and MicroMatrix® Wound Study
Status: Terminated | Type: Observational
Why Stopped: Sponsor Decision
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Winthrop University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CR2017-012
Record Dates: First submitted 2018-08-09; First posted 2018-08-16 (Actual); Results first posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Wounds
Keywords: Wounds; ACell; ACell MicroMatrix®; ACell Cytal® Wound Matrix; Extracellular Matrix; Urinary Bladder Matrix
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Formalin fixed paraffin-embedded wound biopsy tissue.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- ACell Arm: Cytal® Wound Matrix and/or MicroMatrix®
  Cytal® Wound Matrix 1-Layer is composed of porcine-derived extracellular matrix also known as urinary bladder matrix. It is intended for the management of a variety of wounds. The individual device is intended for one time use.
  MicroMatrix® is composed of a porcine-derived extracellular matrix known as urinary bladder matrix and is intended for the management of a variety of wounds. The devices are supplied in particle form in masses up to 1000mg. It is intended for one-time use.
  Interventions: Device: ACell Arm

INTERVENTIONS:
Device: ACell Arm — Cytal® Wound Matrix and/or MicroMatrix®

SUMMARY:
This is an observational study to assess the safety and efficacy of MicroMatrix® alone or in combination with Cytal® Wound Matrix on primary measures of wound healing.

DETAILED DESCRIPTION:
A single-site, prospective, observational clinical study of Cytal® Wound Matrix alone or in combination with MicroMatrix® for the management of wounds. Up to 100 patients with multiple wound types including but not limited to, venous ulcers, diabetic foot ulcers, trauma wounds, and external surgical wounds will be treated either with Cytal® Wound Matrix alone or with Cytal® Wound Matrix and MicroMatrix® for wounds exceeding 3mm in depth. Wound healing efficacy, effect of treatment on patient-reported quality of life, complete wound management, wound-related adverse event, and wound pathology will be measured. The protocol defined patient follow-up is 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has at least one wound that the treating physician determines may be treated with Cytal® with or without MicroMatrix®.
2. Subject is at least 21 years of age.
3. Subject is willing and able to adhere to protocol requirements and agrees to participate in the study program and comply with the study follow-up regimen.
4. Subject or legal representative is willing to provide informed consent.
5. For females of reproductive potential, confirmed negative urine pregnancy test at enrollment.

Exclusion Criteria:

1. Allergy or hypersensitivity to materials in porcine-based study products (per subject report) or personal preference.
2. Subject report of concurrent participation in another clinical trial that involves an investigational drug or device that would interfere with this study.
3. The subject has any condition that, in the Investigator's opinion, would warrant exclusion from the study or prevent the subject from completing the study.
4. The subject's wound shows evidence of infection as determined by the Principal Investigator (which may be indicated by the presence of: elevated WBC, pus, moderate or greater discharge, abnormal odor, or acute osteomyelitis).
5. Wound with exposed organs or hardware.
6. Wound with burn etiology.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from NYU Winthrop Hospital, including the outpatient Wound Healing Center clinic.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Matthews, Study Chair — Integra LifeSciences Corporation
Locations (1):
- NYU Winthrop Hospital, Long Island City, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD to other researchers at this time.

RESULTS

PARTICIPANT FLOW:
Groups:
- ACell Arm: Cytal® Wound Matrix and/or MicroMatrix®
  Cytal® Wound Matrix 1-Layer is composed of porcine-derived extracellular matrix also known as urinary bladder matrix. It is intended for the management of a variety of wounds. The individual device is intended for one time use.
  MicroMatrix® is composed of a porcine-derived extracellular matrix known as urinary bladder matrix and is intended for the management of a variety of wounds. The devices are supplied in particle form in masses up to 1000mg. It is intended for one-time use.
  ACell Arm: Cytal® Wound Matrix and/or MicroMatrix®
Period: Overall Study
Arm/Group | ACell Arm
Started | 37
Completed | 3
Not Completed | 34

BASELINE CHARACTERISTICS:
Arm/Group | ACell Arm
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 24
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Completely Healed Wounds
Description: Assess number of participants with completely healed wounds, defined as 100% epithelialization with no drainage.
Time Frame: Up to 12 weeks
Population: The study was terminated by Sponsor prior to completion, all enrolled subjects did not complete 12 weeks follow-up prior to termination.
Measure: Count of Participants; unit: Participants
Arm/Group | ACell Arm
Number analyzed (Participants) | 23
Participants | 4

2. Primary Outcome: Wound Size Change
Description: Assess wound size at specified intervals. Number of wounds with 40% reduction by week 4, 60% by week 8, and 80% by week 12.
Time Frame: Up to 12 weeks
Population: Data was not collected and outcome measure analysis was not performed.
Arm/Group | ACell Arm
Number analyzed (Participants) | 0

3. Secondary Outcome: Time to Complete Wound Closure
Description: Determine time to complete wound closure using Silhouette Star camera system.
Time Frame: up to 52 week visit (until study completion)
Population: Data was not collected and outcome measure analysis was not performed.
Arm/Group | ACell Arm
Number analyzed (Participants) | 0

4. Secondary Outcome: Wound Characteristics
Description: Identify wound characteristics as determined by granulation tissue quality and presence/quantity of exudate.
Time Frame: up to 52 week visit (until study completion)
Population: Data was not collected and outcome measure analysis was not performed.
Arm/Group | ACell Arm
Number analyzed (Participants) | 0

5. Secondary Outcome: Incidence of Bridging
Description: Bridging to definitive closure or transition to cellular therapy
Time Frame: up to 52 week visit (until study completion)
Population: Data was not collected and outcome measure analysis was not performed.
Arm/Group | ACell Arm
Number analyzed (Participants) | 0

6. Secondary Outcome: Visual Analogue Scale (VAS) for Pain
Description: VAS is a psychometric response scale that measures subjective characteristics or attitudes regarding perceived pain levels from participants. Participants are asked to draw a line on a 10cm horizontal line indicating what their current pain level would be. The distance between the start of the horizontal line to the vertical line is calculated in mm with a higher score (100mm) indicating a greater pain intensity.
Time Frame: Up to 52 week visit (until study completion)
Population: Data was not collected and outcome measure analysis was not performed.
Arm/Group | ACell Arm
Number analyzed (Participants) | 0

7. Secondary Outcome: Wound Quality of Life (W-QOL)
Description: W-QOL is a 17-item Likert style questionnaire that measures 3 subscales in a participant (Body, Psyche, and Everyday to then calculate an overall global score. An overall global score is obtained from averaging all items. Each item is coded with numbers 0 (not at all) to 4 (very much) with a higher score indicating a lower quality of life.
Time Frame: Up to 52 week visit (until study completion)
Population: Data was not collected and outcome measure analysis was not performed.
Arm/Group | ACell Arm
Number analyzed (Participants) | 0

8. Secondary Outcome: Katz Index of Independence in Activities of Daily Living (KATZ ADL)
Description: The Katz ADL is a 6-item questionnaire measuring independence in activities of daily living such as bathing, dressing, toileting, transfers, feeding, and continence. Each item is dichotomized as either having a score of zero (i.e dependence) or one (i.e. independence). An overall score of 6 indicates full function and an overall score of 2 or less indicates severe functional impairment
Time Frame: Up to 52 week visit (until study completion)
Population: Data was not collected and outcome measure analysis was not performed.
Arm/Group | ACell Arm
Number analyzed (Participants) | 0

9. Secondary Outcome: Complete Wound Management
Description: Assess the method of application of products and how it is secured as well as adjunctive treatments and dressing.
Time Frame: up to 52 week visit (until study completion)
Population: Data was not collected and outcome measure analysis was not performed.
Arm/Group | ACell Arm
Number analyzed (Participants) | 0

10. Secondary Outcome: Wound-Related Adverse Events
Description: Number and type of wound-related adverse events as recorded on adverse event case report forms.
Time Frame: up to 52 week visit (until study completion)
Population: Data was not collected and outcome measure analysis was not performed.
Arm/Group | ACell Arm
Number analyzed (Participants) | 0

11. Other Pre Specified Outcome: Direct Product and Care Costs
Description: Measures the direct cost of products
Time Frame: up to 52 week visit (until study completion)
Population: Data was not collected and outcome measure analysis was not performed.
Arm/Group | ACell Arm
Number analyzed (Participants) | 0

12. Other Pre Specified Outcome: Indirect Product and Care Costs
Description: Measures the total of the indirect and incidental costs
Time Frame: up to 52 week visit (until study completion)
Population: Data was not collected and outcome measure analysis was not performed.
Arm/Group | ACell Arm
Number analyzed (Participants) | 0

13. Other Pre Specified Outcome: Return to Work Status
Description: Measures change in "return to work status" and/or "reported work status"
Time Frame: up to 52 week visit (until study completion)
Population: Data was not collected and outcome measure analysis was not performed.
Arm/Group | ACell Arm
Number analyzed (Participants) | 0

14. Other Pre Specified Outcome: Cost Associated With AEs, UADEs and SAEs
Description: Measure frequency of wound specific events, capturing incident specific costs per event.
Time Frame: up to 52 week visit (until study completion)
Population: Data was not collected and outcome measure analysis was not performed.
Arm/Group | ACell Arm
Number analyzed (Participants) | 0

15. Other Pre Specified Outcome: Wound Pathology
Description: Measures the effect of treatment through quantitative analysis
Time Frame: Up to 12 weeks
Population: Data was not collected and outcome measure analysis was not performed.
Arm/Group | ACell Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | ACell Arm
All-Cause Mortality (participants affected / at risk) | 1/37
Serious Adverse Events (participants affected / at risk) | 6/37
Other Adverse Events (participants affected / at risk) | 17/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACell Arm (N=37)
inpatient wound management (General disorders) | 1 (1)
abdominal pain/septic shock (Infections and infestations) | 1 (1)
bacteremia (Infections and infestations) | 1 (1)
discharge at device application site (Infections and infestations) | 1 (1)
urinary tract infection/sepsis (Infections and infestations) | 1 (1)
accidental fall (Musculoskeletal and connective tissue disorders) | 1 (1)
shortness of breath/cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
scheduled surgery and hospitalization (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACell Arm (N=37)
atrial fibrillation (Cardiac disorders) | 1 (1)
bleeding at wound site (General disorders) | 1 (1)
hematoma at device application site (General disorders) | 1 (1)
increase in wound size (General disorders) | 6 (7)
inflammation at device application site (General disorders) | 1 (1)
malaise (General disorders) | 1 (1)
near syncope episode (General disorders) | 1 (1)
pain at application site, discharge at application site (General disorders) | 1 (1)
pain at device application site (excessive or exacerbated) (General disorders) | 1 (1)
cellulitis at device application site (Infections and infestations) | 1 (1)
cellulitis, leg (Infections and infestations) | 1 (1)
conjunctivitis (Infections and infestations) | 1 (1)
osteomyelitis at device application site (Infections and infestations) | 1 (1)
urinary tract infection (Infections and infestations) | 1 (2)
wrist injury (Musculoskeletal and connective tissue disorders) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
burning sensation (Skin and subcutaneous tissue disorders) | 1 (1)
facial rash (Skin and subcutaneous tissue disorders) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 1 (1)
seroma (Skin and subcutaneous tissue disorders) | 3 (4)
skin maceration (Skin and subcutaneous tissue disorders) | 1 (1)
small maculopapular rash (possible reaction to complex wound dressing) (Skin and subcutaneous tissue disorders) | 1 (1)
wound necrosis (Skin and subcutaneous tissue disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Due to early termination, additional primary, secondary, and tertiary endpoint analyses were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/54/NCT03632954/Prot_SAP_000.pdf